CLINICAL TRIAL: NCT03922152
Title: Short-course Accelerated 2D-radiotherapy in Palliative Treatment of Advanced Esophageal Cancer
Brief Title: 2D-radiotherapy in Palliation of Advanced Esophageal Cancer
Acronym: SHARON-2D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Alessio Giuseppe Morganti, Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHARON ESOPHAGUS-2D
Record Dates: First submitted 2019-04-17; First posted 2019-04-19 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Palliative Care
Keywords: palliative care; radiotherapy; pain; quality of life; esophageal cancer
MeSH Terms: conditions — Pain; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Short course radiotherapy (Experimental): The radiotherapy is delivered over 2 days with accelerated hypo-fractionation and 2D-technique.
  Interventions: Radiation: Short course radiotherapy

INTERVENTIONS:
Radiation: Short course radiotherapy — An accelerated hypo-fractionation 2D-radiotherapy is delivered for palliation in patients with advanced esophageal cancer.

SUMMARY:
The study wants to define the efficacy of a short course 2D-radiation therapy in patients with symptomatic advanced esophageal cancer.

DETAILED DESCRIPTION:
The study wants to define the efficacy of a short course accelerated 2D-radiation therapy delivered in twice daily fractions and 2 consecutive days for symptomatic palliation of advanced esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven advanced esophageal cancer
* excluded from curative therapy because of disease stage and/or presence of multiple comorbidities and/or poor performance status
* age > 18 years
* Eastern Cooperative Oncology Group (ECOG) <3

Exclusion Criteria:

* prior radiotherapy to the same region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Assessment of symptoms [odynophagia, chest-back pain, dysphagia, regurgitation] | 1 year
  Symptoms were graded using the IAEA scoring system. Values range from 0 (no symptom) to 4 (severe symptom).

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Acute radiation toxicity] | 1 year
  Acute toxicity after treatment is evaluated with the Radiation Therapy Oncology Group (RTOG) scale. Values range from 0 (no acute toxicity) to 4 (maximum acute toxicity).
Assessment of the Performance Status | 1 year
  Performance Status after the treatment is evaluated according with the Eastern Cooperative Oncology Group (ECOG) score. Values range from 0 (better status) to 5 (worst status).
Assessment of the Overall Survival | 1 year
  Overall Survival is evaluated from the end of radiotherapy to the last date of follow-up. It is calculated in months.

CONTACTS AND LOCATIONS:
Overall Officials: Alessio G. Morganti, MD, Principal Investigator — Radiation Oncology Center, DIMES, University of Bologna, S.Orsola-Malpighi Hospital, Bologna, Italy